CLINICAL TRIAL: NCT05216952
Title: Ulipristal Acetate for Use in Early Pregnancy Loss: A Phase 2 Pilot Feasibility Study
Brief Title: Ulipristal Acetate for Use in Early Pregnancy Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-2315; C21-1493 (Other: UNC Chapel Hill Clinical Research Management)
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Missed Abortion; Anembryonic Pregnancy; Non-Viable Pregnancy
Keywords: Medical management of miscarriage
MeSH Terms: conditions — Abortion, Missed | interventions — ulipristal acetate; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UPA 90mg (Experimental): Participants receive ulipristal acetate 90mg PO followed by self-administration of misoprostol 800mcg vaginally 6 to 18 hours following ulipristal acetate administration.
  Interventions: Drug: Ulipristal Acetate Tablets; Drug: Misoprostol Pill

INTERVENTIONS:
Drug: Ulipristal Acetate Tablets — 90mg (three 30mg tablets) administered orally once
  Other Names: Ella
Drug: Misoprostol Pill — 800mcg (four 200mcg pills) administered vaginally once 6-18 hours following ulipristal acetate
  Other Names: Cytotec

SUMMARY:
The investigators will study the feasibility of using 90mg ulipristal acetate, a selective progesterone receptor agonist, as an adjunct to 800mcg vaginal misoprostol for the medical management of early pregnancy loss. Patients will be followed to assess effective treatment of early pregnancy loss, additional interventions needed, side effects, adverse events and patient acceptability.

DETAILED DESCRIPTION:
Study Background: Early pregnancy loss affects approximately 10% of women throughout their reproductive lives and many women desire medical management of early pregnancy loss. Data from two large randomized controlled trials suggests that pretreatment with mifepristone 200mg, a selective progesterone receptor modulator, prior to administration of misoprostol 800mcg increases effectiveness of medical management of early pregnancy loss and decreases the need for subsequent surgical management. Ulipristal acetate (UPA) is another selective progesterone receptor modulator that may allow for similar priming of the cervix and sensitization of the myometrium to the prostaglandins to improve effectiveness of misoprostol in medical management of early pregnancy loss. Ulipristal acetate is available as a prescription medication through commercial pharmacies. Thus, utilizing UPA plus misoprostol for early pregnancy loss may improve access to patients.

Study Objectives:

Primary Objective:

- To assess if 90mg ulipristal acetate as an adjunct to 800mcg vaginal misoprostol is a feasible method for medical management of early pregnancy loss.

Secondary Objectives:

* To evaluate if participants taking ulipristal acetate plus misoprostol achieve complete resolution of early pregnancy loss.
* To investigate if patients using ulipristal acetate plus misoprostol have side effects or adverse events when used for early pregnancy loss.
* To identify if patients find ulipristal acetate and misoprostol an acceptable treatment for early pregnancy loss.

Study Population: Participants eligible for the study include women over age 18 presenting with a non-viable pregnancy between 5- and 12-weeks gestation or an anembryonic gestation and desiring medical management.

Study Location: All study activities will take place at University of North Carolina-Chapel Hill (UNC). Participants will be recruited from OBGYN clinics following diagnosis of early pregnancy loss on viability scan. All follow up study activities will take place at UNC Chapel Hill Family Planning Clinic.

Study Intervention: Ulipristal acetate is a selective progesterone receptor modulator that is currently FDA approved for the use of emergency contraception. Three 30mg tablets will be administered orally for a total dose of 90mg. Participants will be instructed to self-administer 800mcg of misoprostol 6 to 18 hours after receiving ulipristal acetate as per the standard of care for early pregnancy loss management. Participants will be followed for resolution of their early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older
* English- or Spanish-speaking
* Ultrasound examination showing a non-viable intrauterine pregnancy between 5- and 12-weeks' gestation or anembryonic gestation
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Desire for non-medical management of early pregnancy loss (either expectant management or surgical management)
* Hemodynamically unstable
* Evidence of incomplete or inevitable abortion (due to high efficacy of misoprostol alone)
* Contraindication or allergy to ulipristal acetate or misoprostol (glaucoma, mitral stenosis, sickle cell anemia, chronic glucocorticoid use)
* Evidence of a viable intrauterine pregnancy, ectopic pregnancy, or pregnancy with intrauterine device in place
* Evidence of pelvic infection
* Hemoglobin <9.5g/dL
* Known cardiovascular disease (arrhythmia, cardiac failure, valvular disease, angina)
* Known clotting or bleeding disorder, or on anticoagulation therapy
* Use of the following medications that may influence metabolization of the study medications: barbiturates, bosentan, carbamazepine, felbamate, griseofulvin, oxcarbazepine, phenytoin, rifampin, St. John's Wort, topiramate
* Use of CYP3A4 inhibitors within five elimination half-lives of ulipristal acetate or other strong CYP3A4 inhibitors
* Chronic adrenal failure (risk of acute renal insufficiency)
* Concurrent long-term corticosteroid therapy (risk of acute renal insufficiency)
* Any history of underlying liver disorder, including hepatitis
* Elevation of any or all liver enzymes (alanine aminotransferase, aspartate aminotransferase, total bilirubin) above the upper limit of normal (ULN) at baseline testing prior to enrollment
* A family history of hepatitis or currently living with a person who has been given a diagnosis of hepatitis
* A history of or currently working as a sex worker
* A history of or currently using intravenous (IV) drugs
* A self-reported history of alcohol dependency or abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Hagey, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - University of North Carolina, Chapel Hill - Same Day OBGYN Clinic, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill - Vilcom Center, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill - Weaver Crossing, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill - Hillsborough Medical Office Building, Hillsborough, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, statistical analysis plan and informed consent form will be shared beginning 9 to 36 months following publication of results.
Access Criteria: Following approval from an appropriate review board as described above and execution of a data use/sharing agreement with UNC-Chapel Hill.

RESULTS

PARTICIPANT FLOW:
Groups:
- Ulipristal Acetate (UPA) 90 mg: Participants receive ulipristal acetate 90 mg PO followed by self-administration of misoprostol 800 mcg vaginally 6 to 18 hours following ulipristal acetate administration.
  Ulipristal Acetate Tablets: 90 mg (three 30 mg tablets) administered orally once
  Misoprostol Pill: 800 mcg (four 200 mcg pills) administered vaginally once 6-18 hours following ulipristal acetate
Period: Overall Study
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 34 [33 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Recruited to Study Protocol
Description: Measured as number of participants enrolled in study divided by number of patients screened for participation in study
Time Frame: Baseline
Population: The number of potential participants screened for study eligibility.
Measure: Number; unit: percentage of participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 8
percentage of participants | 37.5

2. Primary Outcome: Percentage of Participants Adherent to Study Protocol
Description: Measured as number of participants self reporting adherence to study intervention of ulipristal acetate followed by misoprostol taken 6-18 hours later divided by number of participants enrolled in study.
Time Frame: From admission until day 3 follow up, +/- 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
percentage of participants | 100

3. Primary Outcome: Percentage of Participants Retained in Study Protocol
Description: Measured as number of participants attending all required study visits (day 0, day 3, day 8, and day 30) divided by number of participants enrolled in study
Time Frame: From admission until day 30 follow up, +/- 7 days
Measure: Number; unit: percentage of participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
percentage of participants | 100

4. Secondary Outcome: Number of Participants With Resolution of Early Pregnancy Loss Following Study Intervention
Description: Absence of gestational sac on transvaginal ultrasound examination on day 3 follow up
Time Frame: From admission until day 3 follow up, +/- 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Number of Participants With Treatment-Related Side Effects
Description: Participant reported side effects based on pre-specified list of common side effects (fatigue, headache, dizziness, chills, nausea, diarrhea, vomiting, severe cramping, and fever) that may occur with medication management of early pregnancy loss.
Time Frame: From admission until day 30 follow up, +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
Participants
  Fatigue | 2
  Headache | 0
  Dizziness | 2
  Chills | 1
  Nausea | 1
  Diarrhea | 0
  Vomiting | 0
  Severe cramping | 1
  Fever | 0

6. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Participant reported adverse events based on pre-specified list (bleeding requiring hospitalization and/or blood transfusion, pelvic infection requiring hospitalization and/or antibiotics) that may occur with medication management of early pregnancy loss.
Time Frame: From admission until day 30 follow up, +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
Participants
  Bleeding requiring hospitalization and/or blood transfusion | 1
  Pelvic infection requiring hospitalization and/or antibiotics | 0
  Other | 0

7. Secondary Outcome: Median Acceptability of Study Intervention
Description: Participant reported ordinal data based on 4 Likert scale questions about acceptability of study intervention with scores ranging from 1-5 (1=Very Unlikely, 2=More Unlikely, 3=Neutral, 4=More Likely, 5=Very Likely). Higher scores indicated more acceptable treatment.
Time Frame: From admission until day 30 follow up, +/- 7 days
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
score on a scale
  Would you use these medications again if you had another miscarriage? | 3 [1 to 5]
  Would you recommend these medications to a friend with a miscarriage? | 4 [3 to 5]
  If possible to take Ulipristal Acetate (UPA) at home, would you be more or less likely to use again? | 4 [3 to 4]
  If possible to take UPA at a different time, would you be more or less likely to use again? | 3 [3 to 4]

8. Other Pre Specified Outcome: Number of Participants Needing Additional Medication for Resolution of Early Pregnancy Loss
Description: Participant reported need for additional dose of misoprostol for resolution of early pregnancy loss.
Time Frame: From admission until day 30 follow up, +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
Participants | 0

9. Other Pre Specified Outcome: Number of Participants Needing Surgical Management for Resolution of Early Pregnancy Loss
Description: Participant reported need for vacuum aspiration for resolution of early pregnancy loss.
Time Frame: From admission until day 30 follow up, +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate (UPA) 90 mg
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, 30 days +/- 7 days.
Arm/Group | Ulipristal Acetate (UPA) 90 mg
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulipristal Acetate (UPA) 90 mg (N=3)
Vaginal Bleeding Requiring Hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulipristal Acetate (UPA) 90 mg (N=3)
Fatigue (General disorders) | 2 (2)
Dizziness (General disorders) | 2 (2)
Chills (Infections and infestations) | 1 (1)
Severe cramping (Reproductive system and breast disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT05216952/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT05216952/ICF_000.pdf